CLINICAL TRIAL: NCT00428142
Title: A Multi-Centre Phase II Trial Investigating the Efficacy and Tolerability of Bortezomib Added to Cyclophosphamide, Vincristine, Prednisone, and Rituximab (BCVP-R) for Patients With Advanced Stage Follicular Non-Hodgkin's Lymphoma Requiring Systemic First-Line Treatment
Brief Title: Bortezomib, Combination Chemotherapy, and Rituximab as First-Line Therapy in Treating Patients With Stage III or Stage IV Follicular Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LY13; CAN-NCIC-LY13; CDR0000527275 (Other: PDQ)
Record Dates: First submitted 2007-01-25; First posted 2007-01-29 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2012-11

CONDITIONS: Lymphoma
Keywords: stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular | interventions — Rituximab; Bortezomib; Cyclophosphamide; Prednisone; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bortezomib + BCVP-R (Experimental): BCVP-R - q 21 days x 4 cycles Bortezomib: 1.3 mg/m2 Days 1 & 8 Cyclophosphamide: 750 mg/m2 IV Day 1 Vincristine: 1.4 mg/m2 IV Day 1 (dose capped at 2 mg) Prednisone: 40 mg/m2 po Days 1-5 Rituximab: 375 mg/m2 IV Day 1
  Interventions: Biological: rituximab; Drug: bortezomib; Drug: cyclophosphamide; Drug: prednisone; Drug: vincristine sulfate

INTERVENTIONS:
Biological: rituximab — 375mg/m2 day 1
Drug: bortezomib — 1.3mg/m2 days 1 & 8
Drug: cyclophosphamide — 750mg/m2 day 1
Drug: prednisone — 40mg/m2 days 1-5
Drug: vincristine sulfate — 1.4mg/m2 day 1 (dose capped at 2mg)

SUMMARY:
RATIONALE: Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as cyclophosphamide, vincristine, and prednisone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Giving bortezomib together with combination chemotherapy and rituximab may kill more cancer cells.

PURPOSE: This phase II trial is studying the side effects and how well giving bortezomib together with combination chemotherapy and rituximab works when given as first-line therapy in treating patients with stage III or stage IV follicular non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess the efficacy of systemic first-line treatment comprising bortezomib, cyclophosphamide, vincristine, prednisone, and rituximab, in terms of complete response rate, in patients with stage III or IV follicular non-Hodgkin's lymphoma.
* Assess the incidence of severe neurotoxicity (defined as grade 3 or 4 neuropathy or neuropathic pain during the first 4 courses of treatment) in patients treated with this regimen.

Secondary

* Assess the overall response rate and response duration in patients treated with this regimen.
* Determine progression-free and overall survival of patients treated with this regimen.
* Evaluate the tolerability and characterize the toxicity profile of this regimen in these patients.
* Assess quality of life, with particular focus on neurotoxicity-related changes, of patients treated with this regimen.

OUTLINE: This is a multicenter, nonrandomized, open-label study.

Patient receive cyclophosphamide IV over 15-45 minutes, vincristine IV over 3-5 seconds and rituximab IV over 1½-6 hours on day 1, oral prednisone daily on days 1-5, and bortezomib IV over 3-5 seconds on days 1 and 8. Treatment repeats every 3 weeks for up to 8 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, at the end of each course of treatment, and on day 42 at the post treatment visit.

After completion of study treatment, patients are followed at 3 and 6 weeks and then every 3-6 months thereafter.

PROJECTED ACCRUAL: A total of 90 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed follicular non-Hodgkin's lymphoma meeting the following criteria:

  * Stage III or IV disease
  * Grade 1, 2, or 3 disease requiring systemic first-line treatment
  * No transformation to diffuse large cell lymphoma
* At least 1 bidimensionally measurable lesion meeting 1 of the following criteria:

  * Lymph nodes > 1.5 cm x 1.0 cm by physical exam or CT scan
  * Other non-nodal lesion ≥ 1.0 cm x 1.0 cm by MRI or CT scan OR ≥ 1.0 cm x 1.0 cm (e.g., skin lesions or nodules) by physical exam
* Must have a medical indication for treatment, as indicated by 1 of the following:

  * Presence of constitutional symptoms that are attributed to lymphoma (e.g., B symptoms, including night sweats, fever, weight loss, fatigue, or pain)
  * Lymphadenopathy that requires treatment based on presence of associated symptoms, potential threat to organ function (e.g., ureteric compromise from retroperitoneal disease), or degree of enlargement (i.e., > 5 cm)
  * Impairment of normal organ function (e.g., impaired hematopoiesis due to marrow involvement by lymphoma or from splenomegaly and hypersplenism)
  * Immune-related complications of lymphoma that require therapy
  * Rate of disease progression for which observation is deemed inappropriate
* No history of any other lymphoproliferative disorder or evidence of transformation to an aggressive histology lymphoma
* No known CNS involvement by lymphoma

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 12 weeks
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Platelet count ≥ 75,000/mm^3*
* Absolute neutrophil count ≥ 1,000/mm^3*
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN
* AST or ALT ≤ 2.5 times ULN (5 times ULN if liver involvement with lymphoma)
* Able (i.e., sufficiently fluent) and willing to complete the quality of life questionnaires in either English or French

  * Inability (illiteracy in English or French, loss of sight, or other equivalent reason) to complete the questionnaires will not make the patient ineligible for the study
* No history of other malignancies, except for the following:

  * Adequately treated nonmelanoma skin cancer
  * Curatively treated in situ cancer of the cervix
  * Ductal carcinoma in situ of the breast (as long as radiation limitation is not exceeded)
  * Other solid tumors curatively treated with no evidence of disease for > 5 years
* No history of allergic reactions attributed to compounds containing boron or mannitol
* No history of an unusual or severe allergic reaction to rituximab or similar agent
* No pre-existing neuropathy ≥ grade 2
* No known HIV infection
* No other serious illness or medical condition that would preclude study participation, including any of the following:

  * Active, uncontrolled bacterial, fungal, or viral infection
  * Significant cardiac dysfunction
  * Cardiovascular disease NOTE: *Exceptions will be allowed for values below these thresholds in patients with marrow involvement by lymphoma or lymphoma-related hypersplenism

PRIOR CONCURRENT THERAPY:

* No prior systemic therapy for lymphoma
* No prior bortezomib, cyclophosphamide, or vincristine
* At least 4 weeks since prior radiotherapy that involved ≤ 25% of functioning bone marrow and recovered

  * Exceptions may be made for low-dose, nonmyelosuppressive radiotherapy or if the irradiated field is not a significant marrow-bearing area
* At least 2 weeks since prior major surgery
* No other concurrent anticancer therapy, investigational agents, corticosteroids (except for physiologic replacement or antiemesis), cytotoxic chemotherapy, or immunotherapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2007-05-01 (Actual); Primary Completion 2011-04 (Actual); Study Completion 2012-01-06 (Actual)

PRIMARY OUTCOMES:
Complete response rate | 5 years
Incidence of severe grade 3 or 4 neurotoxicity or neuropathic pain during the first 4 courses of treatment | 5 years

SECONDARY OUTCOMES:
Overall response rate | 5 years
Response duration in patients with observed responses | 5 years
Time to progression | 5 years
Overall survival | 5 years
Toxicity | 5 years
Quality of life | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Laurie Sehn, Study Chair — British Columbia Cancer Agency; Michael R. Crump, MD, FRCPC, Study Chair — Princess Margaret Hospital, Canada
Locations (19):
- Canada (19):
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA - Fraser Valley Cancer Centre, Surrey, British Columbia
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - BCCA - Vancouver Island Cancer Centre, Victoria, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - The Moncton Hospital, Moncton, New Brunswick
  - QEII Health Sciences Center, Halifax, Nova Scotia
  - Regional Cancer Program of the Hopital Regional, Greater Sudbury, Ontario
  - London Regional Cancer Program, London, Ontario
  - Credit Valley Hospital, Mississauga, Ontario
  - Thunder Bay Regional Health Science Centre, Thunder Bay, Ontario
  - Odette Cancer Centre, Toronto, Ontario
  - Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario
  - Humber River Regional Hospital, Toronto, Ontario
  - Hopital Charles LeMoyne, Greenfield Park, Quebec
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
  - McGill University - Dept. Oncology, Montreal, Quebec
  - CHA-Hopital Du St-Sacrement, Québec, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan

REFERENCES:
- [Result] Sehn LH, Macdonald DA, Rubin SH, et al.: Tolerability and efficacy of bortezomib added to CVP-R for previously untreated advanced stage follicular fymphoma: interim analysis of a phase II study by the NCIC Clinical Trials Group. [Abstract] Blood 112 (11): A-1576, 2008.
- [Result] Sehn LH, MacDonald D, Rubin S, Cantin G, Rubinger M, Lemieux B, Basi S, Imrie K, Gascoyne RD, Sussman J, Chen BE, Djurfeldt M, Shepherd L, Couban S, Crump M. Bortezomib ADDED to R-CVP is safe and effective for previously untreated advanced-stage follicular lymphoma: a phase II study by the National Cancer Institute of Canada Clinical Trials Group. J Clin Oncol. 2011 Sep 1;29(25):3396-401. doi: 10.1200/JCO.2010.33.6594. Epub 2011 Aug 1. PMID 21810681